CLINICAL TRIAL: NCT01882998
Title: PRIMARY HIV PREVENTION IN PREGNANT AND LACTATING UGANDAN WOMEN: A RANDOMIZED TRIAL
Brief Title: Primary HIV Prevention in Pregnant and Lactating Ugandan Women
Acronym: PRIMAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD070767 (NIH); 1R01HD070767-01A1 (NIH)
Record Dates: First submitted 2013-06-17; First posted 2013-06-21 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Primary Prevention of HIV Acquisition
Keywords: HIV and pregnancy; HIV and breastfeeding; Mother-to-child transmission of HIV; Africa; Uganda
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Women-Extended Repeat Testing and Enhanced Counseling (Experimental): Pregnant/breastfeeding women enrolled individually and randomized to the intervention arm will receive extended repeat HIV testing and enhanced counseling at the time of labor and delivery and throughout the lactation period at 3, 6, 12, 18 and 24 months postpartum or until cessation of breastfeeding, whichever occurs first.
  Interventions: Behavioral: Extended repeat HIV testing and enhanced counseling
- Couples-Extended Repeat Testing and Enhanced Counseling (Experimental): Pregnant/breastfeeding women enrolled in couples with their male partners and randomized to the intervention arm will receive extended repeat HIV testing and enhanced counseling at the time of labor and delivery and throughout the lactation period at 3, 6, 12, 18 and 24 months postpartum or until cessation of breastfeeding, whichever occurs first.
  Interventions: Behavioral: Extended repeat HIV testing and enhanced counseling

INTERVENTIONS:
Behavioral: Extended repeat HIV testing and enhanced counseling — Pregnant/breastfeeding women in the intervention arm and their male partners if present will receive extended repeat HIV testing and enhanced counseling around the time of labor and delivery and throughout the breastfeeding period.
  Other Names: ERHTEC

SUMMARY:
This study aims to test the effectiveness of a behavioral intervention aimed at preventing the primary acquisition of HIV by uninfected pregnant and lactating women in Uganda, East Africa where HIV transmission is high. Women who acquire HIV during pregnancy or lactation are at higher risk of adverse health and pregnancy outcomes and their baby is at high risk of acquiring HIV and dying.

Keeping HIV-uninfected women uninfected during pregnancy and lactation is an important component of the global World Health Organization (WHO) strategy to eliminate mother-to-child transmission of HIV but there has been no study to date to assess interventions that can effectively keep these women uninfected.

In this study, the investigators will test the hypotheses that:

1. extended repeat HIV testing and enhanced counseling (ERHTEC) during late pregnancy (>36 weeks) and breastfeeding can increase and sustain risk reduction behaviors and prevent incident STI and HIV infections among HIV-uninfected pregnant women, and
2. that couple HIV testing and counseling (HTC) can further enhance this effect through improved couple communication and emotional and economic support from male partners.

DETAILED DESCRIPTION:
The specific aims of the study are:

* Aim 1: to assess the effect of an extended repeat HIV testing and enhanced counseling (ERHTEC) intervention on sexual risk behavior and sexually transmitted infections (STI) and HIV acquisition in HIV-uninfected pregnant and lactating women enrolled individually
* Aim 2: to assess the effect of ERHTEC on sexual risk behavior and the incidence of STI and HIV in uninfected pregnant and lactating women enrolled with their partner, and
* Aim 3: to assess the costs and estimate the cost-effectiveness of the intervention.

We will conduct a stratified randomized trial of 410 HIV-negative pregnant Ugandan women enrolled individually and 410 HIV-negative pregnant women enrolled with their male partners in Mulago Hospital, Kampala and St Joseph Hospital, Kitgum, Northern Uganda. In each site, 205 women enrolled individually and 205 couples will be randomized to be either retested and counseled for HIV in late pregnancy only (>36 weeks) as per the WHO/Ministry of Health (MOH) recommendation, or to receive ERHTEC throughout pregnancy and breastfeeding.

Individual women and couples randomized to the intervention arm will receive the ERHTEC intervention at 3, 6, 12, and 18 months postpartum. Follow-up will end at 24 months postpartum or 6 weeks after the end of breastfeeding, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Women: 15-49 years old, confirmed HIV negative, confirmed pregnant, living within 30kms /19 miles of hospital, willingness to sign informed consent
* Men: > or = 15 years old, being an established partner of a woman participant, living within 30kms /19 miles of hospital, willingness to sign informed consent

Exclusion Criteria:

* condition requiring hospitalization

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1230 (Actual)
Dates: Start 2013-02; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Frequency of unprotected sex | 27 months
  Self-reported number of unprotected sex episodes among women participants validated by detection of semen (Y chromosome) in vaginal swabs

SECONDARY OUTCOMES:
STI incidence | 27 months
  Incidence of Syphilis, N. gonorrhea, C. trachomatis and T. vaginalis infections among women and men participants
HIV incidence | 27 months
  Incidence of HIV infection among women and men participants
Incidence of recurrent wanted and unwanted pregnancy | 24 months
  Incidence of wanted and unwanted recurrent pregnancy within 24 months of delivery

CONTACTS AND LOCATIONS:
Overall Officials: Jaco Homsy, MD, MPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Result] King R, Bannink F, Mwambi K, Achiro S, Namusoke B, Ajok M, Oweka B, Akot C, Nalubega MG, Adengo M, Namukwaya Z, Homsy J. Primary prevention of HIV among pregnant and lactating women; the neglected PMTCT prong. 7th ICASA Conference, Cape Town, South Africa, 7-11 December 2013. Abstract 2420101.
- [Derived] Bannink Mbazzi F, Namukwaya Z, Amone A, Ojok F, Etima J, Byamugisha J, Katabira E, Fowler MG, Homsy J, King R; PRIMAL Study Team. "[Repeat] testing and counseling is one of the key [services] that the government should continue providing": participants' perceptions on extended repeat HIV testing and enhanced counseling (ERHTEC) for primary HIV prevention in pregnant and lactating women in the PRIMAL study, Uganda. BMC Public Health. 2020 May 15;20(1):694. doi: 10.1186/s12889-020-08738-x. PMID 32414405
- [Derived] Homsy J, King R, Bannink F, Namukwaya Z, Vittinghof E, Amone A, Ojok F, Rukundo G, Amama S, Etima J, Matovu J, Weissglas F, Ojom L, Atim P, Darbes L, Byamugisha J, Rutherford G, Katabira E, Fowler MG; PRIMAL Study Team. Primary HIV prevention in pregnant and lactating Ugandan women: A randomized trial. PLoS One. 2019 Feb 25;14(2):e0212119. doi: 10.1371/journal.pone.0212119. eCollection 2019. PMID 30802277
- See also: Makerere University - Johns Hopkins University Research Collaboration — http://www.mujhu.org